CLINICAL TRIAL: NCT01255696
Title: A Phase 2a, Double-Blind, Placebo Controlled Study of the Efficacy, Safety and Tolerability of 6-weeks Treatment With Varying Methods of ALV003 Administration in Patients With Well-Controlled Celiac Disease
Brief Title: Safety and Efficacy of Varying Methods of ALV003 Administration for the Treatment of Celiac Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alvine Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALV003-1021; 2010-023127-23 (EudraCT Number)
Record Dates: First submitted 2010-12-03; First posted 2010-12-07 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-07

CONDITIONS: Celiac Disease
Keywords: Celiac Disease; Coeliac Disease; Celiac Sprue; Keliakia Disease
MeSH Terms: conditions — Celiac Disease | interventions — ALV003

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALV003 (Experimental): ALV003 is an orally administered mixture of two recombinant proteases (cysteine endoprotease B-isoform 2 and prolyl endopeptidase) engineered to degrade gluten into non-immunogenic fragments, by targeting the glutamine and proline residues common in gluten.
  Interventions: Biological: ALV003
- Placebo (Placebo Comparator): Excipients for ALV003 absent the experimental compounds
  Interventions: Biological: ALV003 placebo

INTERVENTIONS:
Biological: ALV003
  Arms: ALV003
Biological: ALV003 placebo
  Arms: Placebo

SUMMARY:
A phase 2a study to evaluate the safety and efficacy of ALV003 to treat celiac disease.

ELIGIBILITY:
Inclusion Criteria:

* History of biopsy-proven celiac disease
* Adherence to a gluten-free diet
* TG2 antibody negative
* Signed informed consent

Exclusion Criteria:

* Active dermatitis herpetiformis
* History of IgE-mediated reactions to gluten
* Use of specific medications 6 months prior to entry
* History of alcohol abuse or illicit drug use
* Current untreated or GI disease
* Positive pregnancy test
* Received any experimental drug within 14 days of randomization
* Uncontrolled chronic disease or condition
* Uncontrolled complications of celiac disease
* Any medical condition which could adversely affect study participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-11; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Efficacy: Intestinal mucosal morphology | 6 weeks
  Intestinal mucosal morphology - change from baseline to week 6
Safety: Tolerability of ALV003 | 6 weeks
  Safety will be evaluated by collection of adverse events, blood chemistry and blood cell counts

SECONDARY OUTCOMES:
Efficacy: Change in intestinal intraepithelial lymphocyte numbers/phenotype | 6 weeks
  Intestinal intraepithelial lymphocyte numbers/phenotype - change from baseline to week 6
Efficacy: Change in serological markers of celiac disease | 6 weeks
  Serological markers of celiac disease - change from baseline to week 6

CONTACTS AND LOCATIONS:
Overall Officials: Marja-Leena Lähdeaho, MD, Principal Investigator — FINN-MEDI Research Oy; Markku Mäki, MD, PhD, Study Chair — Tampere University
Locations (3):
- Finland (3):
  - Terveystalo Kuopio, Kuopio
  - Oulu Diakonissalaitos (ODL), Oulu
  - FINN-MEDI Research Oy - Clinical Trials Center, Tampere

REFERENCES:
- [Derived] Lahdeaho ML, Kaukinen K, Laurila K, Vuotikka P, Koivurova OP, Karja-Lahdensuu T, Marcantonio A, Adelman DC, Maki M. Glutenase ALV003 attenuates gluten-induced mucosal injury in patients with celiac disease. Gastroenterology. 2014 Jun;146(7):1649-58. doi: 10.1053/j.gastro.2014.02.031. Epub 2014 Feb 25. PMID 24583059